CLINICAL TRIAL: NCT03350321
Title: A Randomized, Open-label, Active-controlled, Parallel-group, Multicenter Study to Investigate the Efficacy and Safety of Oral Molidustat in Comparison to Darbepoetin Alfa in Non-dialysis Subjects With Renal Anemia Who Are Not Treated With Erythropoiesis-Stimulating Agents (ESAs)
Brief Title: A Study of Molidustat for Correction of Renal Anemia in Non-dialysis Subjects
Acronym: MIYABI ND-C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19349
Record Dates: First submitted 2017-11-19; First posted 2017-11-22 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Anemia; Renal Insufficiency, Chronic
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — molidustat; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molidustat (BAY85-3934) (Experimental): Molidustat group
  Interventions: Drug: Molidustat (BAY85-3934)
- Darbepoetin alfa (Active Comparator): Darbepoetin alfa group
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Molidustat (BAY85-3934) — Starting dose of molidustat once daily (OD) will be titrated based on the subject's Hb (Hemoglobin) response
  Arms: Molidustat (BAY85-3934)
Drug: Darbepoetin alfa — Starting dose of darbepoetin alfa once every 2 weeks will be titrated based on the subject's Hb (Hemoglobin) response
  Arms: Darbepoetin alfa

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of molidustat in non-dialysis subjects with renal anemia who are not treated with Erythropoiesis-Stimulating Agents (ESAs).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with estimated glomerular filtration rate (eGFR)< 60 mL/min/1.73m^2 (Chronic kidney disease [CKD] stages 3 to 5)
* Body weight > 40 and ≤ 160 kg at screening
* Male or female subject ≥ 20 years of age at screening
* Not on dialysis and not expected to start dialysis during the study period
* Not treated with ESAs and/or HIF-PH inhibitors within 8 weeks prior to randomization
* Mean of the last 2 central laboratory Hb levels during the screening period must be ≥ 8.0 and < 11.0 g/dL (2 measurements must be taken ≥ 2 days apart and the difference between the 2 measurements must be < 1.2 g/dL) and the last measurements must be taken within 14 days prior to randomization
* Ferritin ≥ 50 ng/mL at screening

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV congestive heart failure
* History of cardio- (cerebro-) vascular events (e.g., unstable angina, myocardial infarction, stroke, pulmonary thromboembolism, and acute limb ischemia) within 6 months prior to randomization
* Sustained and poorly controlled arterial hypertension (defined as systolic BP≥ 180mmHg or diastolic BP ≥ 110mmHg) or hypotension (defined as systolic BP < 90mmHg) at randomization
* Proliferative choroidal or retinal disease, such as neovascular age-related macular degeneration or proliferative diabetic retinopathy requiring invasive treatment (e.g., intraocular injections or laser photocoagulation)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Mean Hb (Hemoglobin) level | From week 30 to 36
Change in hemoglobin level from baseline to the average during the evaluation period | Baseline and week 30 to 36

SECONDARY OUTCOMES:
Responder rate: proportion of responders among the subjects | From week 30 to 36
  Responder is defined as meeting all of the following criteria:
  (i) Mean of the Hb levels in the target range (ii) ≥ 50% of the Hb levels in the target range (iii) No rescue treatment
Rate of rise in Hb (Hemoglobin) level (g/dL/week) | Up to 8 weeks
Rate of rise in Hb (Hemoglobin) level (g/dL/week) | Up to 4 weeks
Proportion of subjects who meet each component of the response | From week 30 to 36
  Response:
  (i) Mean of the Hb levels in the target range (ii) ≥ 50% of the Hb levels in the target range (iii) No rescue treatment
Cumulative proportion of subjects who achieve the lower limit of the target Hb range at least once | Up to 52 weeks
Change in Hb level | Baseline and up to 52 weeks
Hb level | Baseline and up to 52 weeks
Proportion of subjects whose mean hemoglobin level is in the target range | From week 30 to 36
Proportion of subjects whose mean hemoglobin level is above the target range | From week 30 to 36
Proportion of subjects whose mean hemoglobin level is below the target range | From week 30 to 36
Proportion of subjects with hemoglobin levels in the target range | Up to 52 weeks
Proportion of subjects with hemoglobin levels above the target range | Up to 52 weeks
Proportion of subjects with hemoglobin levels below the target range | Up to 52 weeks
Proportion of subjects whose maximum rise in Hb between each consecutive visits is above 0.5 g/dL/week | Up to 52 weeks
  Defined as change in Hb level / duration between two visits (weeks)
Number of participants with serious adverse events | Up to 52 weeks
Maximum concentration (Cmax) | At baseline, week 12, week 24 and week 52
Area under the concentration-time curve (AUC) | At baseline, week 12, week 24 and week 52
EPO (Erythropoietin) serum concentration | At baseline, week 12, week 24 and week 52

CONTACTS AND LOCATIONS:
Locations (61):
- Japan (61):
  - Kainan Hospital, Yatomi, Aichi-ken
  - Seikeikai New Tokyo Heart Clinic, Matsudo, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Saiseikai Matsuyama Hospital, Matsuyama, Ehime
  - Iizuka Hospital, Iizuka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - National Fukuoka-Higashi Medical Center, Koga, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - St.Mary's Hospital, Kurume, Fukuoka
  - Matsunami Health Promotion Clinic, Hashima-gun, Gifu
  - Gifu Prefectural Tajimi Hospital, Tajimi, Gifu
  - Mazda Hospital of Mazda Motor Corporation, Aki-gun, Hiroshima
  - Nippon Kokan Fukuyama Hospital, Fukuyama, Hiroshima
  - Teine Keijinkai Clinic, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - National Hospital Organization Kobe Medical Center, Kobe, Hyōgo
  - National hospital Organization Mito Medical Center, Higashiibaraki, Ibaraki
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - KenAiKai medical corporation Akiyama clinic, Takamatsu, Kagawa-ken
  - Ikeda Hospital, Kanoya, Kagoshima-ken
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Koukan Clinic, Kawasaki, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Arao Municipal Hospital, Arao, Kumamoto
  - Kumamoto Rosai Hospital, Yatsushiro, Kumamoto
  - Uji-Tokushukai Medical Center, Uji, Kyoto
  - JCHO Yokkaichi Hazu Medical Center, Yokkaichi, Mie-ken
  - Japanese Red Cross Ishinomaki Hospital, Ishinomaki, Miyagi
  - Asama Nanroku Komoro Medical Center, Komoro, Nagano
  - Niigata Prefectural Shibata Hospital, Shibata, Niigata
  - Okinawa prefectural Chubu Hospital, Uruma, Okinawa
  - Osaka Saiseikai Senri Hospital, Suita, Osaka
  - Osaka Pref. Saiseikai Tondabayashi Hospital, Tondabayashi, Osaka
  - Kitasato University Medical Center, Kitamoto, Saitama
  - Iwata City Hospital, Iwata, Shizuoka
  - Toshima Hospital, Itabashi-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Showa University Koto Toyosu Hospital, Koto-ku, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Fukui Prefectural Hospital, Fukui
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Asahi University Hospital, Gifu
  - National Hospital Organization Kochi National Hospital, Kochi
  - Nara Prefecture General Medical Center, Nara
  - Kitano Hospital, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Red Cross Hospital, Osaka
  - Nippon Life Hospital, Osaka
  - Chibune Clinic, Osaka
  - Osaka General Medical Center, Osaka
  - Social Corporation Keigakukai Minamiosaka Hospital, Osaka
  - Japanese Red Cross Oita Hospital, Ōita
  - Shizuoka Saiseikai General Hospital, Shizuoka
  - Suruga Clinic, Shizuoka
  - Wakayama Medical University Hospital, Wakayama

REFERENCES:
- [Derived] Yamamoto H, Yamada T, Miyazaki K, Yamashita T, Kato T, Ohara K, Nakamura Y, Akizawa T. Treatment satisfaction with molidustat in CKD-related anemia in non-dialysis patients: a post-hoc analysis of two clinical trials. Clin Exp Nephrol. 2023 Aug;27(8):651-659. doi: 10.1007/s10157-023-02353-x. Epub 2023 Apr 24. PMID 37095342
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Yamamoto H, Taguchi M, Matsuda Y, Iekushi K, Yamada T, Akizawa T. Molidustat for the treatment of renal anaemia in patients with non-dialysis-dependent chronic kidney disease: design and rationale of two phase III studies. BMJ Open. 2019 Jun 14;9(6):e026704. doi: 10.1136/bmjopen-2018-026704. PMID 31203242
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/